CLINICAL TRIAL: NCT01013779
Title: A Phase II Efficacy Study of Chemo-Radiotherapy in PET Stage II and III Merkel Cell Carcinoma of the Skin
Brief Title: Merkel Positron Emission Tomography (PET) Protocol
Acronym: MP3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 09.03; ACTRN12610000480088 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Merkel Cell Carcinoma
Keywords: Merkel Cell Cancer; PET scanning
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Carboplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Experimental): Conventional radical radiotherapy in this trial means that those patients with microscopic disease receive a dose of 50Gy using daily incremental fractions of 2Gy over 25 fractions and those with macroscopic disease receive 54Gy in 27 fractions.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Carboplatin — During radiotherapy: Carboplatin (AUC2) commences on day 1 of radiation and is repeated at weekly intervals on days 8, 15, 22 and 29 (of radiation).
  After radiotherapy: 3 weeks after completing radiotherapy, 3 cycles of 3 weekly carboplatin (AUC4.5) intravenously on day 1.
Drug: Etoposide — After Radiotherapy: 3 weeks after completing the radiation therapy, 3 cycles of 3 weekly etoposide (80mg/M2/day) intravenously days 1-3
Radiation: Radiotherapy — Microscopic Disease: 50Gy delivered in 2Gy doses over 25 fractions
  Macroscopic Disease: 54Gy delivered in 2Gy doses over 27 fractions
  Other Names: RT; Radiation Therapy

SUMMARY:
A Phase II Study designed to evaluate the efficacy of Chemo-Radiotherapy in achieving loco-regional control in patients with Merkel Cell Carcinoma (MCC) of the skin. Patients will undergo PET scans to assist in staging and planning the patient's treatment as well as assessing response at the conclusion of treatment.

ELIGIBILITY:
Inclusion Criteria for Trial Registration:

Patients may be registered on the trial only if they meet all of the following criteria:

* Age 18 years or older
* Written informed consent to participate in the study
* Able to undergo 18-FDG PET scan (no uncontrolled diabetes mellitus or severe claustrophobia).
* Available for follow-up.
* Using adequate contraception if capable of child bearing
* Any Merkel Cell carcinoma confined to the primary and/or nodal sites
* ECOG 0-2.
* Full Blood Count (FBC) should be satisfactory ( Haemoglobin > or equal to 10g/dl, neutrophils > or equal to 2.0 x 109 /l and platelets > or equal to 100 x 109 /l) and renal function (GFR > or equal to 50 ml/min) and hepatic function ( ALT < 5 X upper limit normal, bilirubin < 1.5 X upper limit normal)
* Patients must be able to tolerate protocol treatment

Exclusion Criteria for Registration:

* Previous chemotherapy in the past 5 years or prior radiotherapy to the area of concern
* Unable to comply with treatment protocol eg dementia
* Other malignancy in the past 5 years other than non-melanoma skin cancer.
* Women who are pregnant or lactating.
* Clinical evidence of metastatic disease.
* Immunosuppression from long term steroid use or immunosuppressive drugs.
* Any serious illness or medical condition that precludes the safe administration of the chemotherapy including:

  1. Active infection
  2. Uncontrolled or unstable cardiac disease including unstable angina, myocardial infarction within the last 3 months, and recurrent ventricular arrhythmias

Inclusion Criteria for Treatment Registration:

Patients may proceed to protocol treatment if they meet the following criteria:

* High risk disease with no evidence of distant spread: Biopsy proven MCC with a primary that is > 2cm (T2N0M0= Stage II) and/or regional nodes (any T, N1M0= Stage III); OR Recurrent MCC not previously treated with radiation treatment; Dermal or in-transit metastasis with or without nodes; Occult primary with involved nodes
* Patients who have no metastases on CT or PET scan OR If CT is suggestive of metastases, they must be PET negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Time to loco-regional failure curve | Minimum of 18 months follow up
Incidence of grade 3 and 4 toxicity and incidence of febrile neutropenia | Duration of Radiotherapy treatment

SECONDARY OUTCOMES:
Overall survival and time to distant failure curves | 3 year acturarial curves
Proportion of patients for which PET can influence management. | 12 weeks post Radiotherapy
Positive Predictive Value (PPV) and Negative Predictive Value (NPV) of PET. | 12 weeks post Radiotherapy
Post-treatment PET complete response rate for patients with unresected disease | 12 weeks post Radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Poulsen, Study Chair — Trans Tasman Radiation Oncology Group
Locations (13):
- Australia (13):
  - Campbelltown, Campbelltown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Prince Alfred, Sydney, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Radiation Oncology Services - Mater Centre, Brisbane, Queensland
  - Princess Alexandra Hospital Radiation Oncology, Brisbane, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - Oncology Research Australia, Toowoomba, Queensland
  - Genesis Cancer Care (previously Premion), Tugun, Queensland
  - Geelong Hospital, Geelong, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner, Nedlands, Western Australia

REFERENCES:
- See also: please visit this website for further trial specific information — http://www.trog.com.au